CLINICAL TRIAL: NCT07399223
Title: Comparison of the Metabolomic Effects of Sevoflurane and Desflurane Anesthesia in Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Ahmet Atlas, associate professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hru/25.05.05
Record Dates: First submitted 2026-01-05; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sevoflurane Desflurane; Metabolomic Effect
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane group (Active Comparator)
  Interventions: Procedure: Sevoflurane
- desflurane group (Active Comparator)
  Interventions: Procedure: Desflurane

INTERVENTIONS:
Procedure: Sevoflurane — This group will be operated on under sevoflurane.
  Arms: sevoflurane group
Procedure: Desflurane — This group will be operated on under desflurane.
  Arms: desflurane group

SUMMARY:
Analytical techniques used in metabolomic studies include nuclear magnetic resonance (NMR) spectroscopy and mass spectrometry (MS). The study will involve comparing the metabolomic profiles of patients receiving sevoflurane and desflurane during surgery to identify any differences in metabolic pathways affected by the two anaesthetic techniques. Metabolomic profiles are generated using spectroscopic and spectrometric techniques such as high-field NMR and MS, as well as separation techniques.

DETAILED DESCRIPTION:
Our study will include 100 patients undergoing laparoscopic cholecystectomy surgery, divided into two groups. Patients aged 18-65 years with an ASA I-II classification, who will undergo laparoscopic cholecystectomy surgery, have no active infection, and have a body mass index (BMI) <35, and who agree to participate in the study, will be intubated after standard anaesthetic induction (propofol, rocuronium, fentanyl) and intubated. The first sample will be taken from the finger immediately after the inhalation anaesthetic (sevoflurane, desflurane) reaches 1 minimal alveolar concentration (MAC) level. The second sample will be taken after the surgical procedure is completed and the inhalation anaesthesia is discontinued. The samples will be taken from the patients' fingertips and absorbed onto Guthrie paper. Statistical analysis will be performed on the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy surgery who have no active infection, Body mass index (BMI)<35, Aged 18-65, ASA I-II, and who agree to participate in the study

Exclusion Criteria:

* Individuals over 65 years of age ASA 3-4 patients Individuals with a body mass index (BMI) >35 Smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
amino acid metabolism | 12 weeks
Our primary outcome measure will be the effect of both inhalation anaesthetics on amino acid metabolism. | 12 weeks

IPD SHARING:
Plan to Share IPD: No